CLINICAL TRIAL: NCT06146348
Title: Adapting and Testing a Deimplementation Program in the Intensive Care Unit
Brief Title: Deimplementing CXR After CVC (DRAUP) in the ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Enyo Ablordeppey, Assoc Prof of Anesthesiology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202312113; 5K01HL161026-02 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Implementation Science; Behavior and Behavior Mechanisms
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CVC confirmed by DRAUP (Experimental): new mode of CVC confirmation for correct location and excluding pneumothorax
  Interventions: Behavioral: adapted DRAUP strategy bundle
- CVC confirmed by CXR (Experimental): traditional mode of CVC confirmation for correct location and excluding pneumothorax
  Interventions: Behavioral: adapted DRAUP strategy bundle

INTERVENTIONS:
Behavioral: adapted DRAUP strategy bundle — DRAUP deimplementation strategy bundle includes: 1) education and training, 2) supervision and in-person decision support, and 3) audit and feedback to target capability. Opportunity is addressed by 4) algorithm development and 5) organizational support. Finally, 6) facilitators and 7) planned adaptation after interval program assessment address the motivations needed to change behavior.

SUMMARY:
This study proposes adapting and testing an innovative, behavioral theory-driven deimplementation program called DRAUP in two intensive care units for proof of concept and support that the program can help providers and hospital organizations address context determinants of deimplementation. Study data will be used to optimize the intervention for a subsequent larger trials.

DETAILED DESCRIPTION:
There are millions of critically ill patients annually who require imaging confirmation after central venous catheter insertion. Emerging literature demonstrates that ultrasound is a faster alternative to historical chest xray, thus serving as the ideal confirmation for catheter use. When able to confirm catheter position, ultrasound decreases the number of unnecessary chest radiographs, cumulative resources (technologist, radiologist, equipment), and patient care delays. However, providers are not adopting this practice. Previously, we developed and initiated a successful evidence-based deimplementation program for ultrasound in lieu of chest xray called DRAUP in the Emergency Department. We now move to adapt the deimplementation bundle in the new environment of the Intensive Care Unit (ICU) with hopeful continued success.

In experiment 1, qualitative analysis will be employ a systematic approach to DRAUP component refinement dosed to the unique context of the Intensive Care Unit and implementation outcomes as well as cost will be evaluated. In experiment 3, mixed methods will be used to evaluate the mechanism of impact of the refined program in the new environment.

ELIGIBILITY:
-Measure the effectiveness and cost effectiveness of DRAUP on discontinuation of CXRs

Inclusion Criteria for DRAUP training:

(1) ICU faculty, fellows, senior residents (post graduate year 3) and advanced practice practitioners

* ICU inclusion for DRAUP program:
* Availability of ultrasound machines with archiving capability (DICOM)
* A minimum of 100 supradiaphragmatic CVC insertions annually in adult patients (age >18)
* Capacity to access digital archiving (PICOM)
* Patient inclusion for DRAUP program:
* supradiaphragmatic CVC placed
* Patient exclusion for DRAUP program:
* severe instability (cardiac arrest, severe shock) where CVC would be used without CXR,
* level 1 trauma;
* burn patients with no viable skin surface for imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DRAUP in | 24 months
  Deadoption of CXR after US guided CVC confirmation

SECONDARY OUTCOMES:
Fidelity | 24 months
  Percentage of DRAUP non-adherence

CONTACTS AND LOCATIONS:
Overall Officials: Enyo Ablordeppey, MD MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing upon request
Supporting Information: Study Protocol